CLINICAL TRIAL: NCT07267819
Title: The Efficacy of Xeomin as a Prophylactic Therapy for Migraine in Patients With Traumatic Brain Injuries (TBIs) Versus Anomalous Health Incidents (AHIs)
Brief Title: Efficacy of Xeomin for Migraines in Patients With Traumatic Brain Injuries vs. Anomalous Health Incidents
Status: Recruiting | Type: Observational
Sponsor: Uniformed Services University of the Health Sciences (U.S. Federal Agency)
Responsible Party: Principal Investigator, David Brody, Professor of Neurology, Uniformed Services University, Uniformed Services University of the Health Sciences
Other Study IDs: USUHS.2025-154
Record Dates: First submitted 2025-09-11; First posted 2025-12-05 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Migraine; Traumatic Brain Injury; Anomalous Health Incidents
Keywords: Anomalous health incident; Traumatic brain injury; Headache; Migraine; Botulinumtoxin
MeSH Terms: conditions — Migraine Disorders; Brain Injuries, Traumatic; Headache | interventions — incobotulinumtoxinA

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- TBI Cohort: Patients with a history of Traumatic Brain Injury (TBI) receiving Xeomin treatments for migraine management. The anticipated number of participants is 40.
  Interventions: Drug: Xeomin (incobotulinumtoxinA)
- AHI Cohort: Patients with a history of Anomalous Health Incidents (AHI) receiving Xeomin treatments for migraine management. The anticipated number of participants is 20.
  Interventions: Drug: Xeomin (incobotulinumtoxinA)

INTERVENTIONS:
Drug: Xeomin (incobotulinumtoxinA) — Patients receive their scheduled Xeomin treatment as prescribed by their physician as part of their standard of care. The treatment protocol (dosage, injection sites, etc.) will be documented.

SUMMARY:
This cohort study aims to compare the efficacy of Xeomin injections for migraine management in patients with a history of Traumatic Brain Injury (TBI) versus those with a history of Anomalous Health Incidents (AHI). The study will be conducted at the National Intrepid Center of Excellence (NICOE) in Bethesda, MD. The primary objective is to determine if Xeomin injections result in different outcomes for migraine management between TBI and AHI patients. This is a combined retrospective and prospective cohort study design. Patients scheduled for Xeomin treatments will be categorized into TBI and AHI groups. For the prospective cohort, participants will complete a baseline questionnaire, receive their scheduled Xeomin treatment, and participate in follow-up interviews at 4-6 weeks and 10-12 weeks post-treatment. For the retrospective cohort, similar information will be acquired from existing records. Statistical analysis will compare migraine characteristics and treatment responses between the two groups. All data will be de-identified to protect patient privacy.

DETAILED DESCRIPTION:
Headaches with migraine-like characteristics are a common sequelae of traumatic brain injury (TBI)¹-⁴ and Havana syndrome, otherwise known as anomalous health incidents (AHIs).⁵,⁶ In TBI patients, direct biomechanical forces lead to cellular injury and neuroinflammation, contributing to post-traumatic headaches. Specifically, the disruption of trigeminovascular pathways and the release of inflammatory mediators, such as calcitonin gene-related peptide (CGRP), are implicated in the pathophysiology of post-traumatic migraines. Furthermore, the presence of comorbid conditions, such as post-concussive syndrome, can exacerbate headache symptoms and complicate treatment strategies.⁷ Though the migraine-like headaches in patients with AHI are clinically similar to those seen in patients with mTBI, the absence of clear structural damage on conventional neuroimaging in many AHI cases raises questions about the underlying mechanisms.⁸,⁹ Theories involving unknown exposure and subsequent disruption of white matter function have been proposed. Some analyses suggest that the symptoms of AHI could result from the disruption of neuroimmune and neurotransmission mechanisms similar to those affected in patients with TBI.¹⁰,¹¹

Managing post-traumatic headaches involves a multidisciplinary approach including behavioral therapy, physical therapy, oral medications, injectable medications, and interventional procedures. Essentially, these headaches can be treated similarly to the primary headache disorder they resemble.¹² Thus, the post-traumatic migraine can be treated in the acute setting with triptans, NSAIDs, ergot alkaloids, antiemetics, and other therapeutics.¹³,¹⁴ For chronic management, options include beta-blockers, tricyclic antidepressants, CGRP-targeting agents, anti-seizure medications, and many other medications.¹²,¹⁵ Onabotulinum toxin A (OBA) and other medications in the class of botulinum toxins have been particularly effective at reducing the overall frequency and duration of migraines in patients with TBIs,¹⁶,¹⁷ as well as non-TBI-related migraines. OBA results in a blockade of neural stimulation by inhibiting the release of neurotransmitters at the presynaptic terminal.¹⁸,¹⁹ It's thought to reduce the exocytosis of pain mediators (substance P, CGRP) from sensory neurons by cleaving SNAP25.²⁰,²¹ This effect is temporary due to the formation of new synapses, thus patients have to return for repeat injections every 10-12 weeks. Additionally, the number of units of OBA can be optimized to the patient's level of pain during each treatment.

There is limited literature on managing post-AHI headache disorders, but recent experience indicates that using multidisciplinary approaches similar to those used for TBI-related headache disorders may be appropriate.⁶ OBA, and more specifically incobotulinum toxin A (Xeomin brand) has therefore been a commonly used treatment modality in these patient populations in the Military Health System. Many individuals with AHIs from other branches of the government are treated in the MHS though the Secretarial Designee program.

While AHI symptoms might share pathophysiological characteristics with TBIs, there's limited research on Xeomin injections' characteristics in TBI vs. AHI patients, such as treatment frequency and efficacy. This study aims to quantify these similarities and differences in migraine management with Xeomin, potentially improving our understanding of this treatment modality. Migraines can disrupt home, work, and social activities, and treatment can be especially difficult in AHI patients who face limited effective treatment options that are evidence-based, and unique diagnostic challenges. By comparing Xeomin's efficacy in both groups, this study could reveal crucial differences in treatment response, leading to more personalized and effective therapies that align with a holistic healthcare model in medicine. The findings could inform clinical guidelines and improve migraine management in TBI and AHI patients, ultimately reducing the healthcare burden. This research is essential for addressing AHI patients' unmet needs and advancing migraine treatment understanding.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Able to provide written consent in English
* An employee of the US Government, or an adult family member of a US Government employee
* Have received Xeomin treatment to prevent migraine related to TBI or AHI at a Military Treatment Facility or other US Medical Facility
* Able to participate in at least 80% of the assessments
* A US Citizen and not a dual national of the country where you are currently located

Exclusion Criteria:

* Prisoner
* Decisionally impaired and unable to provide informed consent
* Non-US citizen

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Employees of the US Government, or adult family members of US Government employees, receiving Xeomin treatment for migraine headache following either TBI or AHI.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-08-05 (Actual); Primary Completion 2028-06-06 (Estimated); Study Completion 2028-06-06 (Estimated)

PRIMARY OUTCOMES:
Percent Change in Migraine Headache Intensity from Baseline to Peak Effect (4 weeks post-treatment) and to wearing off (12 weeks post-treatment). | Baseline, 4 weeks post-treatment, and 12 weeks post-treatment.
  Comparison between TBI and AHI groups in the percent change of migraine headache intensity. Intensity is assessed using a 0-10 Numeric Rating Scale (NRS) in response to the question, "How painful were the migraine headaches typically at their worst (0-10)?". For this scale, 0 indicates 'no pain' and 10 indicates the 'worst imaginable pain,' where a higher score signifies a worse outcome. The change is measured from baseline ("Before you started Xeomin treatments") to peak effect ("When your Xeomin was at its peak effect").
Percent Change in Migraine Headache Frequency from Baseline to Peak Effect (4 weeks post-treatment) and to wearing off (12 weeks post-treatment). | Baseline, 4 weeks post-treatment, and 12 weeks post-treatment.
  Comparison between TBI and AHI groups in the percent change of migraine headache frequency. Frequency is defined as the total number of migraine headaches in a typical week, as reported on a patient questionnaire. The minimum value for this count is 0, and a higher number indicates a worse outcome. The change is measured from baseline to the time of the treatment's peak effects.
Percent Change in Headache Impact Test (HIT-6) Score from Baseline to Peak Effect (4 weeks post-treatment) and to wearing off (12 weeks post-treatment). | Baseline, 4 weeks post-treatment, and 12 weeks post-treatment.
  Comparison between TBI and AHI groups in the percent change in the Headache Impact Test (HIT-6) score. The HIT-6 is a 6-item questionnaire assessing the impact of headaches on daily life. Patient responses ("Never," "Rarely," "Sometimes," "Very Often," "Always") are converted to a numerical score. The total score ranges from 36 to 78, where a higher score indicates a more severe headache impact, representing a worse outcome. The change is measured from baseline to the time of the treatment's peak effects

SECONDARY OUTCOMES:
Duration of Xeomin Effectiveness. | Up to 12 weeks post-treatment.
  Comparison between TBI and AHI groups regarding the timeline of Xeomin effectiveness, including time to onset of effects and duration of benefits.

CONTACTS AND LOCATIONS:
Locations (1):
- National Intrepid Center of Excellence (NICOE), Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
The study protocol specifies that there are no data sharing or data use agreements in place for this research. The data collected is intended for internal analysis by authorized research personnel only. While de-identified, aggregate results may be published, the consent form assures participants that their individual data will not be shared in any way that would identify them.

REFERENCES:
- [Background] Klein SK, Brown CB, Ostrowski-Delahanty S, Bruckman D, Victorio MC. Identifying Migraine Phenotype Post Traumatic Headache (MPTH) to Guide Overall Recovery From Traumatic Brain Injury. J Child Neurol. 2022 Jun 3:8830738221100327. doi: 10.1177/08830738221100327. Online ahead of print. PMID 35656769
- [Background] Erickson JC. Treatment outcomes of chronic post-traumatic headaches after mild head trauma in US soldiers: an observational study. Headache. 2011 Jun;51(6):932-44. doi: 10.1111/j.1526-4610.2011.01909.x. Epub 2011 May 17. PMID 21592097
- [Background] Becker WJ. Acute Migraine Treatment. Continuum (Minneap Minn). 2015 Aug;21(4 Headache):953-72. doi: 10.1212/CON.0000000000000192. PMID 26252584
- [Background] Pringsheim T, Becker WJ. Triptans for symptomatic treatment of migraine headache. BMJ. 2014 Apr 7;348:g2285. doi: 10.1136/bmj.g2285. No abstract available. PMID 24711666
- [Background] Theeler B, Lucas S, Riechers RG 2nd, Ruff RL. Post-traumatic headaches in civilians and military personnel: a comparative, clinical review. Headache. 2013 Jun;53(6):881-900. doi: 10.1111/head.12123. PMID 23721236
- [Background] Chacko TP, Toole JT, Morris MC, Page J, Forsten RD, Barrett JP, Reinhard MJ, Brewster RC, Costanzo ME, Broderick G. A regulatory pathway model of neuropsychological disruption in Havana syndrome. Front Psychiatry. 2023 Oct 27;14:1180929. doi: 10.3389/fpsyt.2023.1180929. eCollection 2023. PMID 37965360
- [Background] Aristi G, Kamintsky L, Ross M, Bowen C, Calkin C, Friedman A, Hashmi JA. Symptoms reported by Canadians posted in Havana are linked with reduced white matter fibre density. Brain Commun. 2022 Mar 7;4(2):fcac053. doi: 10.1093/braincomms/fcac053. eCollection 2022. PMID 35505689
- [Background] Pierpaoli C, Nayak A, Hafiz R, Irfanoglu MO, Chen G, Taylor P, Hallett M, Hoa M, Pham D, Chou YY, Moses AD, van der Merwe AJ, Lippa SM, Brewer CC, Zalewski CK, Zampieri C, Turtzo LC, Shahim P, Chan L; NIH AHI Intramural Research Program Team; Moore B, Stamps L, Flynn S, Fontana J, Tata S, Lo J, Fernandez MA, Lori-Joseph A, Matsubara J, Goldberg J, Nguyen TD, Sasson N, Lely J, Smith B, King KA, Chisholm J, Christensen J, Magone MT, Cousineau-Krieger C, French LM, Yonter S, Attaripour S, Lai C. Neuroimaging Findings in US Government Personnel and Their Family Members Involved in Anomalous Health Incidents. JAMA. 2024 Apr 2;331(13):1122-1134. doi: 10.1001/jama.2024.2424. PMID 38497822
- [Background] Swanson RL 2nd, Hampton S, Green-McKenzie J, Diaz-Arrastia R, Grady MS, Verma R, Biester R, Duda D, Wolf RL, Smith DH. Neurological Manifestations Among US Government Personnel Reporting Directional Audible and Sensory Phenomena in Havana, Cuba. JAMA. 2018 Mar 20;319(11):1125-1133. doi: 10.1001/jama.2018.1742. PMID 29450484
- [Background] Ruff RL, Blake K. Pathophysiological links between traumatic brain injury and post-traumatic headaches. F1000Res. 2016 Aug 31;5:F1000 Faculty Rev-2116. doi: 10.12688/f1000research.9017.1. eCollection 2016. PMID 27635228
- [Background] National Academies of Sciences, Engineering, and Medicine; Division on Engineering and Physical Sciences; Health and Medicine Division; Standing Committee to Advise the Department of State on Unexplained Health Effects on U.S. Government Employees and Their Families at Overseas Embassies; Pavlin JA, Relman DA, editors. An Assessment of Illness in U.S. Government Employees and Their Families at Overseas Embassies. Washington (DC): National Academies Press (US); 2020 Dec 5. Available from http://www.ncbi.nlm.nih.gov/books/NBK566407/ PMID 33411434
- [Background] Asadi-Pooya AA. Havana syndrome: a scoping review of the existing literature. Rev Environ Health. 2022 Aug 15;38(4):655-661. doi: 10.1515/reveh-2021-0182. Print 2023 Dec 15. PMID 35962646
- [Background] Ashina H, Porreca F, Anderson T, Amin FM, Ashina M, Schytz HW, Dodick DW. Post-traumatic headache: epidemiology and pathophysiological insights. Nat Rev Neurol. 2019 Oct;15(10):607-617. doi: 10.1038/s41582-019-0243-8. Epub 2019 Sep 16. PMID 31527806
- [Background] Lucas S, Hoffman JM, Bell KR, Dikmen S. A prospective study of prevalence and characterization of headache following mild traumatic brain injury. Cephalalgia. 2014 Feb;34(2):93-102. doi: 10.1177/0333102413499645. Epub 2013 Aug 6. PMID 23921798
- [Background] Hoffman JM, Lucas S, Dikmen S, Temkin N. Clinical Perspectives on Headache After Traumatic Brain Injury. PM R. 2020 Oct;12(10):967-974. doi: 10.1002/pmrj.12338. Epub 2020 Mar 2. PMID 32003524
- [Background] Walker WC, Seel RT, Curtiss G, Warden DL. Headache after moderate and severe traumatic brain injury: a longitudinal analysis. Arch Phys Med Rehabil. 2005 Sep;86(9):1793-800. doi: 10.1016/j.apmr.2004.12.042. PMID 16181945

DOCUMENTS (3):
  • Study Protocol (2025-06-05): https://cdn.clinicaltrials.gov/large-docs/19/NCT07267819/Prot_000.pdf
  • Statistical Analysis Plan (2025-06-05): https://cdn.clinicaltrials.gov/large-docs/19/NCT07267819/SAP_001.pdf
  • Informed Consent Form (2025-06-05): https://cdn.clinicaltrials.gov/large-docs/19/NCT07267819/ICF_002.pdf